CLINICAL TRIAL: NCT07261384
Title: "Investigation of the Effects of Individually Tailored Physiotherapy Approaches on Pain, Fatigue, and Physical Function in Individuals With Migraine: A Randomized Controlled Trial"
Brief Title: "Personalized Physiotherapy for Migraine: Effects on Pain, Fatigue, and Physical Function"
Acronym: TIP-MIG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ikra Hatice Dinc, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10333602-050.04-291274
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Migraine
Keywords: Migraine; Fatigue; Pain; Physical Function; Individualized Physical Therapy
MeSH Terms: conditions — Migraine Disorders; Fatigue; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Structured Physiotherapy Intervention (Experimental): Participants will receive a personalized, structured physiotherapy program including manual therapy, cervical spine stabilization exercises, vestibular rehabilitation exercises, and pain neuroscience education. The intervention will be delivered by a licensed physiotherapist twice weekly for 8 weeks.
  The manual therapy will include component, applied according to individual patient needs to reduce pain, improve mobility, and modulate neuromuscular control.
  The cervical spine stabilization exercises will target deep neck flexors and cervical postural muscles to improve neuromuscular control, endurance, and motor coordination.
  The vestibular rehabilitation component will include gaze stabilization, habituation, and balance exercises tailored to migraine-related vestibular symptoms.
  The PNE program will consist of structured individual education sessions focusing on pain neurobiology, central sensitization, and self-management strategies.
  Participants will attend supervised physio
  Interventions: Other: Personalized Structured Physiotherapy Intervention
- Standard Treatment (Active Comparator): Participants will continue their routine migraine care, including any pharmacological treatment. During the 8-week study period, they will receive only two 40-minute Pain Neuroscience Education sessions. No additional physiotherapy or exercise interventions.
  Interventions: Other: Standard Treatment

INTERVENTIONS:
Other: Personalized Structured Physiotherapy Intervention — The manual therapy will include component, applied according to individual patient needs to reduce pain, improve mobility, and modulate neuromuscular control.
  The cervical spine stabilization exercises will target deep neck flexors and cervical postural muscles to improve neuromuscular control, endurance, and motor coordination.
  The vestibular rehabilitation component will include gaze stabilization, habituation, and balance exercises tailored to migraine-related vestibular symptoms.
  The PNE program will consist of structured individual education sessions focusing on pain neurobiology, central sensitization, and self-management strategies.
  Participants will attend supervised physiotherapy sessions twice weekly for 8 weeks, complemented by a personalized home exercise program. All components will be delivered by a licensed physiotherapist.
  Arms: Personalized Structured Physiotherapy Intervention
Other: Standard Treatment — Participants continue routine care including medications prescribed by their physician. Only two 40-minute Pain Neuroscience Education sessions over 8 weeks. No physiotherapy or exercise intervention provided.
  Arms: Standard Treatment

SUMMARY:
Migraine is a prevalent neurological disorder associated with pain, fatigue, and reduced physical function. The aim of this randomized controlled trial is to examine the effects of a personalized and structured physiotherapy program-including cervical spine stabilization exercises, vestibular rehabilitation, and pain neuroscience education-on pain intensity, fatigue, and functional outcomes in individuals with migraine. Participants will be randomly allocated to an intervention group receiving personalized physiotherapy or a control group receiving standard physiotherapy care. Outcomes will be assessed at baseline, post-intervention, and follow-up.

DETAILED DESCRIPTION:
Migraine is a disabling primary headache disorder characterized by recurrent attacks and frequently accompanied by cervical musculoskeletal dysfunction, vestibular symptoms, and altered pain processing mechanisms. Current evidence suggests that physiotherapy interventions targeting manual therapy, cervical stabilization, vestibular function, and pain neuroscience education may positively influence migration-related outcomes; However, studies combining these components in a personalized treatment model are limited.

This randomized controlled trial aims to investigate the effectiveness of a personalized structured physiotherapy program designed specifically for individuals with migraine. The interventions will include manual therapy, cervical spine stabilization exercises, vestibular rehabilitation strategies, and pain neuroscience education delivered by a physiotherapist. The control group will receive only pain neuroscience education.

Primary outcomes will include pain intensity and frequency. Secondary outcomes will include fatigue, disability level, cervical function, physical performance, and patient-reported functional limitations. Assessments will be conducted at baseline, immediately post-intervention, and during a follow-up period. The findings are expected to contribute to evidence-based physiotherapy approaches for migraine management.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 55 years

  * Diagnosed with migraine according to the International Classification of Headache Disorders - 3rd edition (ICHD-3) criteria
  * Experiencing 2-8 migraine attacks per month in the last 3 months
  * Able to participate in an 8-week physiotherapy intervention program
  * Able to understand instructions and provide written informed consent
  * Stable medication use for migraine for at least 1 month prior to participation (no changes planned during study period)

Exclusion Criteria:

* • Presence of other primary headache disorders (cluster headache, tension-type headache as primary diagnosis, etc.)

  * Neurological diseases (epilepsy, stroke, multiple sclerosis)
  * Vestibular disorders unrelated to migraine
  * Cervical radiculopathy, myelopathy, or severe cervical spine pathology
  * History of neck surgery or significant cervical trauma
  * Severe musculoskeletal conditions affecting posture or cervical function
  * Pregnancy or breastfeeding
  * Participation in another clinical trial within the last 3 months
  * Inability to attend intervention sessions or complete outcome assessments

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (VAS) | Baseline, Week 8
  Pain intensity will be assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain). Measurements will be taken at baseline, and at the completion of the 8-week intervention.

SECONDARY OUTCOMES:
Pain Frequency (MIDAS A Question) | Baseline and Week 8
  Pain frequency will be assessed using Question A of the Migraine Disability Assessment Questionnaire (MIDAS), which evaluates the number of headache days over the previous 3 months.
Fatigue (Modified Fatigue Impact Scale - MFIS) | Baseline and Week 8
  Fatigue levels will be measured using the Modified Fatigue Impact Scale (MFIS), which evaluates physical, cognitive, and psychosocial aspects of fatigue.
Migraine Disability (MIDAS Total Score) | Baseline and Week 8
  Migraine-related disability will be assessed with the MIDAS total score, which quantifies the impact of migraine on daily activities over the past 3 months.
Quality of Life (Headache Impact Test - HIT-6) | Baseline and Week 8
  Quality of life will be evaluated using the HIT-6 questionnaire, which measures headache-related impact on daily functioning.
Craniovertebral Angle (Forward Head Posture) | Baseline and Week 8
  Forward head posture will be assessed by measuring the craniovertebral angle using a goniometer, with smaller angles indicating more pronounced forward head posture.
Cervical Range of Motion | Baseline and Week 8
  Cervical mobility (flexion, extension, lateral flexion, rotation) will be measured with a goniometer to assess changes in cervical spine range of motion.
Deep Cervical Flexor Muscle Performance | Baseline and Week 8
  Deep cervical flexor endurance and activation will be assessed using the Stabilizer Pressure Biofeedback Unit during cranio-cervical flexion tasks.
Trigger Point Tenderness / Pressure Pain Threshold | Baseline and Week 8
  Assessment with Manuel compression.
Neck Pain Intensity (VAS) | Baseline, Week 8
  Neck pain intensity will be measured using a 0-10 Visual Analog Scale (VAS) to assess changes over time.
Dizziness Handicap (DHI) | Baseline and Week 8
  Vestibular disability will be assessed with the Dizziness Handicap Inventory (DHI), evaluating functional, emotional, and physical impacts of dizziness.
Balance (Mini-BESTest) | Baseline and Week 8
  Balance performance will be evaluated using the Mini-Balance Evaluation Systems Test (Mini-BESTest), which assesses dynamic balance and postural control.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan Binali Yıldırım Univercity, Medicine Faculty, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The dataset contains sensitive clinical information, and sharing is not planned. Only aggregated results will be available upon publication.